CLINICAL TRIAL: NCT05728203
Title: Audiologic Assessment of Call Center Operators
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya yasser abdelrahman, Principle investigator, Assiut University
Other Study IDs: Audiologic Assessment
Record Dates: First submitted 2023-02-04; First posted 2023-02-15 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Hearing Disorders
MeSH Terms: conditions — Hearing Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Early detection of hearing affection in call center operators
2. Study the effect of this type of noise on the auditory brainstem response.

DETAILED DESCRIPTION:
Occupational noise-induced hearing loss (ONIHL) is a common occupational disease as it is estimated that 1.3 billion people were suffering of hearing loss due to noise exposure. Worldwide, occupational noise exposure is responsible for 16% of cases of disabling hearing loss in adults Commonly, hearing loss interferes with communication and can hinder personal attention and cognition. Older people with mild hearing loss have a twofold increased risk of dementia, whereas those with severe hearing loss have a fivefold increased risk of dementia.

In the last years there was increase in the number of new forms of workplaces, such as call centers. In accordance with the British Health and Safety Executive, a call center is defined as a work environment where all basic employee's tasks are completed simultaneously by phone and on PC. The very first call centers appeared in Europe in Sweden, in the mid-70's of the last century. The last decade brought rapid development of call centers proven by 10percent growth in employment in this sector between 2002and 2007.

Sources of noise occurring in offices can be divided into four categories:

* human activity (for example: noise created by walking people, phone calls including speaker systems),
* office equipment (for example: computers, printers, copy machines, faxes , ringing phones , net devices, mobile headsets),
* building indoor installations (for example: ventilation , heating system and air condition system-HVAC.hydraulic and lift systems),
* outdoor noise (most often a result of traffic).

There are many factors that have impact on indoor noise level such as outside area noise ,neighbor workers from the side as well as from the upper and lower levels activity and finally ,the call center technical equipment, The loudest systems with regard to the last one are ventilation and air condition, in accordance to research , the level of background noise is not high (54-60db) and should not be considered to be a threat towards health ;however, due to focusing employee's involuntary attention on information delivered by noise ,it should be seen as an annoying factor.

To minimize negative auditory health effects on workers in call centers, it is important to assess, and diagnose early occupational hearing loss (OHL) and tinnitus among them. As, early reporting, diagnosis, and intervention can limit the severity of, OHL as it is mostly irreversible. To our knowledge no local previous studies were done in this area.

ELIGIBILITY:
Inclusion Criteria:

* Active working workers in call centers with minimum exposure 2year.
* Had no previous auditory problems.
* Their ages between [18-50] years old working at call centers from 6-12hours/day,5-6days a week.

Exclusion Criteria:

1. evidence of systemic illness [ cardiovascular, renal and diabetes]
2. previous history of hearing loss and tinnitus before working at the call center.
3. History of noise, ototoxic drugs and chemotherapy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Active working workers in call centers with minimum exposure 2year.
  * Had no previous auditory problems.
  * Their ages between [18-50] years old working at call centers from 6-12hours/day,5-6days a week.
Sampling Method: Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Audiologic assessment of call center operators | through study completion, an average 2 years
  By using of audiometer to assess hearing loss and using of auditory brainstem response to assess effect of this type of noise on hearing

CONTACTS AND LOCATIONS:
Overall Officials: Eman A Sayed, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pawlaczyk-Luszczynska M, Dudarewicz A, Zamojska-Daniszewska M, Zaborowski K, Rutkowska-Kaczmarek P. Noise exposure and hearing status among call center operators. Noise Health. 2018 Sep-Oct;20(96):178-189. doi: 10.4103/nah.NAH_11_18. PMID 30516171